CLINICAL TRIAL: NCT03418012
Title: Effect of History-indicated Early Treatment With Cervical Pessary Versus Expectant Management Treatment With Rescue Cerclage in Cases With Cervical Shortening in Singleton Pregnancies at High-risk for sPTB on Children's Long-term Outcome
Brief Title: Prevention of sPTB With Early Cervical Pessary Treatment in Women at High Risk for PTB
Acronym: Prometheus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bürgerhospital Frankfurt (Other)
Responsible Party: Principal Investigator, Ioannis Kyvernitakis, Associate Professor, Bürgerhospital Frankfurt
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BHFKIK2018P
Record Dates: First submitted 2018-01-23; First posted 2018-01-31 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-05

CONDITIONS: Preterm Birth; Premature Birth
Keywords: Cervical Pessary; Short Cervix; Recurrent Preterm Birth; history of cervical surgery; history of conisation
MeSH Terms: conditions — Premature Birth | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: parallel groups:
  * Controll group with management as usual
  * Pessary group with insertion of cervical pessary at 12+0-16+0 weeks of gestation
Masking Description: due to the nature of the intervention (placement of a cervical pessary) a masking is not possible
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cervical Pessary-Group (Experimental): Cervical Pessary Group: placement of the cervical pessary (non-invasive) at enrolment including a transvaginal ultrasound to verify its correct fit. Removal of the cervical pessary (non-invasive) in a regular preventive examination at WoG 37
  Interventions: Device: cervical pessary
- Control-Group (Other): Control-Group women receive management as usual; i.e. expectant management with interventions only in terms of a tertiary prevention of PTB according to guidelines for premature rupture of membranes, premature labour or other pregnancy complications
  Interventions: Other: Control-Group

INTERVENTIONS:
Device: cervical pessary — Intervention: Device: Cervical pessary: After Having excluded a vaginal infection insertion of the cervical pessary (silicone ring) directly after enrollment. After insertion verification of correct fit of the cervical pessary by transvaginal ultrasound. Removal of the pessary at 37+0 weeks of gestation, or before if any unexpected event occurs. Except for the insertion of the pessary the obstetrical management during the remainder of the pregnancy will be usual management.
  Other Names: Arabin Cervical Pessary
  Arms: Cervical Pessary-Group
Other: Control-Group — Intervention: Other: expectant management: expectant management is usual care; interventions only in terms of a tertiary prevention of PTB according to guidelines for premature rupture of membranes, premature labour or other pregnancy complications
  Arms: Control-Group

SUMMARY:
Prevention of preterm birth (PTB) is a key factor for a positive short-term and long-term outcome of the newborn children as mortality and morbidity are inversely related to gestational age at delivery. Consequently every week of prolonged pregnancy will have a tremendous effect concerning the outcome of the new-borns, subsequently for their parents and society as well.

The proposed RCT aims to evaluate the impact of a preventive pessary treatment on the prevention of preterm birth in women with a singleton pregnancy who are at high risk of spontaneous preterm birth (sPTB) due to a history of at least one previous preterm delivery and/or a history of previous cervical surgery. In accordance with the results by "van´t Hooft et al. 2016" an approximately 20% higher percentage of children's long-term survival without neurodevelopmental disability is expected for the pessary group in comparison with usual management (=control group) on basis of a reduction of prematurity < 34 week of gestation (WoG).

The primary outcome measure for the effect of the pessary treatment in comparison to expectant management will be the children's long-term survival (3yrs) without neurodevelopmental disability. Secondary endpoints assess the impact of a preventive pessary placement on the prevention of preterm birth and its resulting risk on mortality and morbidity for the neonates.

DETAILED DESCRIPTION:
The "Prometheus Trial" is a prospective, multicentre, multinational, open-label, randomised, controlled clinical trial in parallel groups.

Up to now the risk factor previous PTB has only been investigated in randomised controlled trials (RCTs) for 17-hydroxyprogesterone caproate (17-OHPC) which is not available in most european countries or in RCTs where the risk factor previous PTB was combined with the risk factor cervical shortening.

Looking at the evidence of therapeutic effectiveness of vaginal progesterone these risk factors should be addressed separately. Vaginal progesterone proved to be ineffective in the prevention of recurrent PTB but effectively reduced PTB in women with a short cervix.

For cervical pessary therapy there is up to now only one cohort analysis for the combined risk factors available proving the placement of a cervical pessary to be as effective as cerclage or treatment with 200 mg vaginal progesterone in reducing preterm birth rate.

The risk factor 'history of at least one cold knife conisation' for PTB was up to now only addressed in a pilot study investigating the effect of pessary treatment in asymptomatic women with a singleton pregnancy along with a short sonographic cervix and it suggested a beneficial effect on the prolongation of the pregnancy.

In approximately 1/3 of pregnancies leading to PTB cervical shortening develops. Here the placement of a cervical pessary is a good therapeutic option. For this risk factor good evidence is available for cervical pessary treatment in singleton and twin pregnancies. This is the first RCT aiming to investigate the impact of a preventive cervical pessary therapy for the prevention of recurrent PTB in women with a history of PTB and/or history of at least one conisation.

Furthermore this RCT is a part of the first worldwide prospective metaanalysis in the medicine Global Obstetrics Network "http://www.globalobstetricsnetwork.org/projects/". The primary outcome "Children´s survival without neurodevelopmental disability at the age of 3 years" measures the long-time outcome of the intervention according to the CROWN criteria.

Cervical pessary treatment is a non-invasive, well-tolerated and cost-effective treatment option which could be easily implemented in daily practice if it proves to have a preventive effect of PTB. This especially applies for developing countries, where for example serial cervix length measurements to detect cervical shortening are not feasible.

Statistics:

The primary statistical aim is to compare the primary combined outcome "long-term survival without neuro-developmental disability at 3 years follow up" between the two treatment groups with a two-sided chi-square test. In general, statistical comparisons will be two-sided and use appropriate tests according to the scale of the outcome. A multivariate logistic regression will be fitted to control for possible confounders. Relative risks and 95% confidence interval as well as adjusted odds ratios will be calculated for the binary outcomes. Statistical significance will be accepted in all cases with a p≤0.05.

The main statistical evaluation will be performed at two time points.

1. The complete data set for the secondary endpoints will be available after the last women enrolled in this study has delivered her neonate, so the analysis of these outcome parameter will be done right after this event.
2. The primary outcome will be evaluated 3 years after the last woman enrolled in this study has delivered her neonate.

A descriptive analysis by preterm birth will be carried out calculating means and medians for quantitative variables and proportions with 95% confidence intervals for categorical variables.

Additionally an explorative subgroup analysis of the study collective will be performed comparing the efficacy of the cervical pessary treatment in women with a normal cervical length at 12 -16 weeks of gestation and in women who have developed a cervical shortening (< 25 mm) as an additional risk factor.

A drop out rate of up to 25% for the primary endpoint is expected due to the long follow-up time (3 years) of the study; but it is not expected to have lost data for the secondary endpoints because for these parameters the study has a short follow-up time till time to birth only.

An interim analysis shall be conducted on key safety parameters after birth of 150 neonates: the following safety endpoints will be assessed by a one-sided test with alpha=1%

* on level of the neonates: rate of preterm birth, time to birth, birth weight, death, neonatal morbidity, harm of intervention
* and on the maternal level: rate of hospitalisation for threatened preterm labour < 32 weeks, rate of PRoM <32 weeks, rate of infection / inflammation, rate of physical or psychological intolerance to pessary, rate of severe adverse reaction (SAR) / severe adverse event (SAE), death.

The trial will be terminated as negative if a disadvantage for the pessary-treatment can be found in one of these tests. To guarantee a high safety level the significance level is chosen more conservatively than in a Bonferroni correction. All analysis will be carried out with SPSS® version 19.0 or later ("IBM Company SPSS Inc." Headquarters, Chicago, Illinois. USA) and R version 3.2.3 or later (R Foundation for Statistical Computing, Vienna, Austria).

Methods against bias:

* all women will be randomly allocated to the cervical pessary group or the control-group in a 1:1 ratio. The randomization sequence is computer generated with variable block sizes using a web-based electronic case report form (e-CRF) (Online-Software Castor is a fully Good Clinical Practice compliant system) stratified for centers. The allocation code will be disclosed after the patient´s initials will be confirmed. The investigators or the trial coordinator will not have access to the randomization sequence.
* Exclusion criteria were chosen to ensure an equal risk distribution for pregnancy complications and fetal morbidity / mortality rate for both study groups.
* The study is open label since masking the intervention is not possible. Investigator training: All investigators should be trained in pessary application and cerclage placement. Quality protocols should be submitted according to the "Clara-Angela Foundation" -requirements for pessary placement.

Outcome assessors will be blinded to the interventions. Group allocations will base on an intention to treat basis with a per protocol allocation as sensitivity analysis.

The study will be registered and the study protocol is available. Outcome measures meet the core-outcome set for the evaluation of interventions to prevent PTB published by the CROWN-initiative.

ELIGIBILITY:
Inclusion Criteria:

* Women with a singleton pregnancy and a history of at least one previous preterm delivery before 34+0 weeks and/or a history of at least one previous cervical surgery
* 12+0 - 16+0 weeks of gestation at time of randomization
* only women with minimum age of 18 and capable of giving consent

Exclusion Criteria:

* major fetal abnormalities
* uterine malformation, placenta previa totalis
* Cerclage prior to randomization
* At randomisation: active vaginal bleeding and/or spontaneous rupture of membranes and/or painful regular uterine contractions
* silicone allergy
* current participation in other RCT

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — only pregnant woman (singleton gestation)
Enrollment: 310 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Children's survival without neurodevelopmental disability at the age of 3 years | assessment of the newborn at age of 3 years (corrected age for prematurity)
  * mortality rate will be recorded
  * neurodevelopmental disability will be assessed by the Ages & Stages questionnaire and by medical examination at 3 years of age (corrected age for prematurity)

SECONDARY OUTCOMES:
rate of preterm birth | randomisation till birth, maximum 25 weeks
  rate of delivery before weeks of gestation: 36+6 / 33+6 / 31+6 / 29+6 / 27+6
time till birth | days from randomisation till birth, maximum 30 weeks
  time span from enrollment till birth
birth weight of the neonate | at birth
  birth weight of the neonate in grams recorded at hospital
Fetal or neonatal death | at birth, first 24 hours after birth
  death of the neonate before birth /within first 24 hours
Need (days) for neonatal special care unit | birth till discharge from hospital, recorded for at least first 48 hrs after birth
  Number of days the neonate is transferred to ICU for medical interventions other than supervision
neonatal morbidity | birth till discharge from hospital, recorded for at least first 48 hrs after birth
  rate of major adverse neonatal outcomes: Intraventricular Haemorrhage III-IV, Retinopathy of prematurity, Respiratory Distress Syndrome II-IV, Need for ventilation > 72 h, Necrotising enterocolitis, Proven or suspected sepsis (antibiotics >5 days)
harm from intervention | birth till discharge from hospital, recorded for at least first 48 hrs after birth
  recording any harm of the neonate deriving from the cervical pessary
maternal death | enrollment till discharge from hospital, recorded for at least first 48 hrs after birth
  rate of maternal death due to pregnancy/birth
rate of significant maternal adverse events | enrollment till discharge from hospital, recorded for at least first 48 hrs after birth
  rate of : heavy bleeding, cervical tear due to pessary placement, uterine rupture
infection/inflammation | enrollment till discharge from hospital, recorded for at least first 48 hrs after birth
  rate of maternal infection and/or inflammation during pregnancy / birth
physical or psychological intolerance to pessary | time from placement of cervical pessary at enrollment till removal of cervical pessary at WoG 37, maximum 25 weeks
  rate of maternal physical or psychological intolerance to pessary during pregnancy
Hospitalisation for threatened preterm labour before 31+6 weeks | randomization till birth, maximum 20 weeks
  Hospitalisation for threatened preterm labour before 31+6 weeks: recording of days of hospitalisation and tocolytic treatment: type / days / dose
premature rupture of membranes (PRoM) before 31+6 weeks | randomization till birth, maximum 20 weeks
  rate of women with premature rupture of membranes (PRoM) before 31+6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ioannis Kyvernitakis, MD, PhD, Study Director — Asklepios Clinic Barmbek
Locations (9):
- University of Adelaide, Adelaide, Australia
- Germany (5):
  - Charité - Universitätsmedizin, Berlin
  - Vivantes Klinikum im Friedrichshain, Berlin
  - Universitätsklinikum Frankfurt, Frankfurt
  - Asklepios Kliniken Krankenhaus Barmbeck, Hamburg
  - Universitätsklinikum des Saarlandes, Homburg
- Greece (2):
  - University Hospital of Athens, Athens
  - Medical School of Aristotle-University of Thessaloniki, Thessaloniki
- Vall d'Hebron University Hospital, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abdel-Aleem H, Shaaban OM, Abdel-Aleem MA, Aboelfadle Mohamed A. Cervical pessary for preventing preterm birth in singleton pregnancies. Cochrane Database Syst Rev. 2022 Dec 1;12(12):CD014508. doi: 10.1002/14651858.CD014508. PMID 36453699

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-29): https://cdn.clinicaltrials.gov/large-docs/12/NCT03418012/Prot_SAP_000.pdf